CLINICAL TRIAL: NCT04842552
Title: The Effect of Hydralazine on the Early Stage of Alzheimer's Disease: A Randomized Clinical Trial
Brief Title: Effect of Hydralazine on Alzheimer's Disease
Acronym: EHSAN
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Sadoughi University of Medical Sciences and Health Services (Other)
Collaborators: National Institute for Medical Research Development (NIMAD) (Unknown); McMaster University (Other)
Responsible Party: Principal Investigator, Masoud Mirzaei, Professor, Shahid Sadoughi University of Medical Sciences and Health Services
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRCT20200711048075N1
Record Dates: First submitted 2021-04-05; First posted 2021-04-13 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-12

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer Disease; Hydralazine; Early stage; Olfactory sense
MeSH Terms: conditions — Alzheimer Disease; Anosmia | interventions — Hydralazine

STUDY DESIGN:
Intervention Model Description: Two arms will be randomly allocated to either hydralazine hydrochloride 25mg TDS or placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Hydralazine hydrochloride was imported directly from a global supplier, packed in 90 tablet bottles with a specific batch number for drug and placebo not revealed to any of the above parties.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Hydralazine hydrochloride 25mg (Active Comparator): Hydralazine hydrochloride (25mg tablets) every eight hours (TDS)
  Interventions: Drug: Hydralazine hydrochloride 25mg tablets
- Placebo (Placebo Comparator): Placebo tablets (identical in shape to the active comparator) every eight hours (TDS)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hydralazine hydrochloride 25mg tablets — Hydralazine hydrochloride 25mg tablets three time daily for 365 days (one year)
  Arms: Hydralazine hydrochloride 25mg
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
It has been recently discovered that the FDA-approved drug, hydralazine, has anti-neurodegenerative efficacy based on three intriguing observations. hydralazine; 1) activates the Nrf2 pathway that controls more than 200 antioxidant proteins, 2) rejuvenates mitochondria and increases their respiration capacity and adenosine triphosphate production, 3) activates autophagy which has pathophysiological roles such as intracellular aggregate clearance. There is an emerging agreement that autophagy-lysosome defects occur early in the pathogenesis of Alzheimer's disease (AD). Nrf2 is another pathway known to be impaired in the hippocampus of AD patients who need antioxidant protection the most. Rejuvenation of mitochondria is crucial for fighting AD, as neuronal cells need more energy to afford activation of pathways such as autophagy and Nrf2. The prime objective of this application is to conduct a randomized clinical trial to assess the efficacy of hydralazine in early-stage AD patients who take one of the acetylcholinesterase inhibitor (AChEI) donepezil, rivastigmine, or galantamine.

DETAILED DESCRIPTION:
Study aim:

1. Determination and comparison of the effect of 75mg (25mg TDS) hydralazine vs. placebo in patients with mild to moderate Alzheimer's disease.
2. Development of an electronic Case Report Form (CRF) and push notification system to remind patients (and/or caregivers) of drug intake to improve drug intake adherence and reduce follow-up losses.
3. Evaluation of the prognostic accuracy of olfactory tests to predict the changes in cognition and performance of patients with mild to moderate Alzheimer's disease.

Design:

This is a phase III, triple-blind, parallel double-armed randomized clinical trial with an allocation ratio of 1-1 to the intervention and placebo arms. This trial will be conducted on 424 randomly selected patients using random permuted blocks.

Settings and conduct:

All patients who are identified as potentially eligible by the supporting neurologists and psychiatrists will be referred to Adineh Clinic to evaluate their cognitive function, assess for inclusion and exclusion criteria and obtain informed consent. The two arms of the study are hydralazine 75mg (25mg three times per day) or hydralazine placebo. A follow-up evaluation will continue for one year after drug administration. The participants, outcome assessors, researchers, and data analyzers will be blinded to the study arms.

Participants/Inclusion and exclusion criteria:

patients over the age of 49 and over who are diagnosed with mild to moderate AD will be included in this study; dementia patients with etiologies other than AD (i.e. vascular dementia) will not be included.

Intervention groups:

The two arms of the study are Hydralazine 75mg (25mg three times per day) or Hydralazine placebo.

Main outcome variables:

Various cognitive and function tests for patients and caregivers, olfactory tests, biochemistry as well as drug side effects will be assessed regularly over the period of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Diagnoses of Alzheimer's disease according to the National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria.
* Presence of a caregiver (friend or relative) who can assume responsibility for medication administrations, accompany the patient to all visits, and rate patient's condition.
* Written informed consent form from both the patient (or surrogate) and caregiver.
* A Mini-Mental State Examination score between 12 and 26 inclusive.
* Prescription of donepezil (5-10mg/d), rivastigmine (3-6mg/d), galantamine or galantamine ER (8-16mg/d) for a minimum of 4 weeks prior to randomization.
* Agreement not to take hydralazine.
* Age 49 and over.

Exclusion Criteria:

* Non-Alzheimer primary dementia diagnosis (e.g., vascular dementia, Lewy body dementia, frontotemporal dementia, vitamin B-12 deficiency, hypothyroidism).
* Diagnosis of any of the following conditions; major depression, delirium, alcohol or psychoactive substance abuse or dependency, schizophrenia, or delusional disorder as defined by Diagnostic and Statistical Manual (DSM)-IV.
* Diagnosis of systemic illnesses that would interfere with participation in the study or decrease the life expectancy to less than one year.
* Currently being treated with hydralazine or a history of intolerance to oral therapy with hydralazine
* Any intravenous treatment for heart failure, except IV furosemide (e.g. IV inotropes, pressors, nitrates or nesiritide) at the time of screening.
* Systolic blood pressure <100 mmHg, reversible etiology of acute heart failure such as myocarditis, acute myocardial infarction-over the past 4 weeks, arrhythmia and existence of pacing device (Acute myocardial infarction is defined as symptoms and major electrocardiogram (ECG) changes (i.e., ST segment elevations), and arrhythmia includes unstable heart rates above 120/min or below 50/min).
* Existence of severe congenital heart disease (such as uncorrected tetralogy of fallot or transposition of the aorta) and severe aortic or mitral stenosis or severe rheumatic mitral regurgitation.
* Concurrent use of phosphodiesterase type 5 (PDE5) inhibitors (e.g. Viagra, Etc.)
* Cardiac revascularization within the last 3 months or likelihood of requiring coronary revascularization within the study period. eGFR (Glomerular Filtration Rate) < 15ml/min/1.73m2, or on regular dialysis, or planned dialysis within the study period.

Min Age: 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Estimated)
Dates: Start 2021-08-02 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-12-20 (Estimated)

PRIMARY OUTCOMES:
The progression of of Alzheimer's disease | Three months after recruitment.
  The progression of of Alzheimer's disease in the hydralazine-treated group compared to placebo-treated using the Alzheimer's Disease Assessment Scale-Cognitive Sub-scale inventory
The progression of of Alzheimer's disease | Six months after recruitment.
  The progression of of Alzheimer's disease in the hydralazine-treated group compared to placebo-treated using the Alzheimer's Disease Assessment Scale-Cognitive Sub-scale inventory
The progression of of Alzheimer's disease | Nine months after recruitment.
  The progression of of Alzheimer's disease in the hydralazine-treated group compared to placebo-treated using the Alzheimer's Disease Assessment Scale-Cognitive Sub-scale inventory
The progression of of Alzheimer's disease | Twelve months after recruitment.
  The progression of of Alzheimer's disease in the hydralazine-treated group compared to placebo-treated using the Alzheimer's Disease Assessment Scale-Cognitive Sub-scale inventory

SECONDARY OUTCOMES:
Function of patients with Alzheimer's disease | Three months after recruitment
  Changes in the function of patients with Alzheimer's disease in the hydralazine-treated group compared to placebo- treated using Lawton Activity of Daily Living Scale
Function of patients with Alzheimer's disease | Six months after recruitment
  Changes in the function of patients with Alzheimer's disease in the hydralazine-treated group compared to placebo- treated using Lawton Activity of Daily Living Scale
Function of patients with Alzheimer's disease | Nine months after recruitment
  Changes in the function of patients with Alzheimer's disease in the hydralazine-treated group compared to placebo- treated using Lawton Activity of Daily Living Scale
Function of patients with Alzheimer's disease | Twelve months after recruitment
  Changes in the function of patients with Alzheimer's disease in the hydralazine-treated group compared to placebo- treated using Lawton Activity of Daily Living Scale
Cognition of patients with Alzheimer's disease | Three months after recruitment
  Changes in the cognition of the patients with Alzheimer's disease in the hydralazine-treated group compared to placebo-treated using Mini Mental State Examination
Cognition of patients with Alzheimer's disease | Six months after recruitment
  Changes in the cognition of the patients with Alzheimer's disease in the hydralazine-treated group compared to placebo-treated using Mini Mental State Examination
Cognition of patients with Alzheimer's disease | Nine months after recruitment
  Changes in the cognition of the patients with Alzheimer's disease in the hydralazine-treated group compared to placebo-treated using Mini Mental State Examination
Cognition of patients with Alzheimer's disease | Twelve months after recruitment
  Changes in the cognition of the patients with Alzheimer's disease in the hydralazine-treated group compared to placebo-treated using Mini Mental State Examination
Behavior of patients with Alzheimer's disease | Three months after recruitment
  Changes in the behaviour of the patients with Alzheimer's disease in the hydralazine-treated group compared to placebo-treated using Nero-Psychiatry Inventory
Behavior of patients with Alzheimer's disease | Six months after recruitment
  Changes in the behaviour of the patients with Alzheimer's disease in the hydralazine-treated group compared to placebo-treated using Nero-Psychiatry Inventory
Behavior of patients with Alzheimer's disease | Nine months after recruitment
  Changes in the behaviour of the patients with Alzheimer's disease in the hydralazine-treated group compared to placebo-treated using Nero-Psychiatry Inventory
Behavior of patients with Alzheimer's disease | Twelve months after recruitment
  Changes in the behaviour of the patients with Alzheimer's disease in the hydralazine-treated group compared to placebo-treated using Nero-Psychiatry Inventory
Caregiver's spent time | Three months after recruitment
  Changes in caregiver's spent time for the patients in the hydralazine-treated group compare to placebo using Caregiver Activity Scale
Caregiver's spent time | Six months after recruitment
  Changes in caregiver's spent time for the patients in the hydralazine-treated group compare to placebo using Caregiver Activity Scale
Caregiver's spent time | Nine months after recruitment
  Changes in caregiver's spent time for the patients in the hydralazine-treated group compare to placebo using Caregiver Activity Scale
Caregiver's spent time | Twelve months after recruitment
  Changes in caregiver's spent time for the patients in the hydralazine-treated group compare to placebo using Caregiver Activity Scale
Olfactory sense | Three months after recruitment
  the changes in the olfactory sense in the hydralazine-treated group compare to placebo using 'peanut butter smelling test'
Olfactory sense | Six months after recruitment
  the changes in the olfactory sense in the hydralazine-treated group compare to placebo using 'peanut butter smelling test'
Olfactory sense | Nine months after recruitment
  the changes in the olfactory sense in the hydralazine-treated group compare to placebo using 'peanut butter smelling test'
Olfactory sense | Twelve months after recruitment
  the changes in the olfactory sense in the hydralazine-treated group compare to placebo using 'peanut butter smelling test'
Drug side effects | Daily records in the provided notebook and reported three month after recruitment. Urgent matter can be reported any time to the provided hotline.
  The side effects of hydralazine-treated group compare to placebo-treated
Drug side effects | Daily records in the provided notebook and reported six month after recruitment. Urgent matter can be reported any time to the provided hotline.
  The side effects of hydralazine-treated group compare to placebo-treated
Drug side effects | Daily records in the provided notebook and reported nine month after recruitment. Urgent matter can be reported any time to the provided hotline.
  The side effects of hydralazine-treated group compare to placebo-treated
Drug side effects | Daily records in the provided notebook and reported twelve month after recruitment. Urgent matter can be reported any time to the provided hotline.
  The side effects of hydralazine-treated group compare to placebo-treated

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Mirzaei, PhD, Study Chair — Shahid Sadoughi University of Medical Sciences
Locations (1):
- Adineh Health Centre, Yazd, Iran

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data (IPD) sharing plan will be decided according to the upcoming requests and the ethics committee approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Informed consent form will be shared after recruitment started. CSR and SAP will be shared after recruitment phase was concluded. Study Protocol will be shared after publication.
Access Criteria: All requests should be forwarded to the study email address and agreed by the investigators' committee subject to the ethics committee approval.
URL: http://ehsan-study.com

REFERENCES:
- See also: The EHSAN study website — http://ehsan-study.com
- Available data/document: Informed Consent Form — http://ehsan-study.com — All requests should be submitted to the contact us/about at the study website or study.ehsan@gmail.com
- Available data/document: Clinical Study Report — http://ehsan-study.com — All requests should be submitted to the contact us/about at the study website or study.ehsan@gmail.com
- Available data/document: Study Protocol — http://ehsan-study.com — All requests should be submitted to the contact us/about at the study website or study.ehsan@gmail.com
- Available data/document: Statistical Analysis Plan — http://ehsan-study.com — All requests should be submitted to the contact us/about at the study website or study.ehsan@gmail.com